CLINICAL TRIAL: NCT06368583
Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' and Providers' Experience During Neuraxial Labour Analgesia. A Prospective Patient-centered Multidisciplinary Quality Improvement Study. (PAS-EDU-NLA)
Brief Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' and Providers' Experience During Neuraxial Labour Analgesia
Acronym: PAS-EDU-NLA
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24-05
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Well-Being, Psychological
Keywords: patient experience; neuraxial analgesia; labour epidural
MeSH Terms: conditions — Psychological Well-Being | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vaginal delivery with neuraxial analgesia: Patients who have a vaginal delivery with neuraxial analgesia.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patients will be interviewed by the research team to learn about their experience of vaginal delivery with neuraxial analgesia
  Other Names: Interview questions

SUMMARY:
During the process of labour and delivery, patients may experience a wide range of events in a short time frame. This study focuses on exploring these experiences and aims to incorporate the improvements from these experiences so that in future, the expectations of patients delivering can be met as much as possible. Since every patient and encounter is unique, they might have a variety of experiences, be it during the labour epidural placement or during the delivery of the baby. Our study aims to explore the patients' perspective and learn about their preferences, concerns and suggestions regarding their experience and to then use this information to enhance the quality of future anesthesia care during labour and delivery.

Patients who underwent labour and delivery and received labour epidural for pain management will be approached the day following the delivery, while their recollection of their experience is still fresh, and given the opportunity to participate in the study which will involve the completion of a questionnaire as well as an interview lasting approximately 20-25 minutes. In addition to interviewing the patients, the study will also involve several interviews of the obstetricians, anesthesiologists, and nurses with the goals of seeing how the patients' experiences compare to the providers' perspective of the care they are delivering. Following the gathering of this information and identification of potential improvements in current practice, a follow up study will be performed aiming to implement changes and improve the quality of anesthesia care during labour and delivery.

DETAILED DESCRIPTION:
About 85-90% of parturient receive labour epidural as a method of pain management for labour and delivery. Various factors play a role in requesting an epidural. Proper patient counseling and education before Labour Epidural Analgesia (LEA) alleviates patient's anxiety and also ensures safety. There are a limited number of studies that have explored the experience of the patient while undergoing LEA and labour and delivery, and even fewer that have focused on the patients' perspective that is used to educate health care professionals on how to improve the quality of anesthesia care during LEA. This study embraces the patient perspective to guide quality improvement in labour and delivery.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older
* ASA Physical Classification Score II or III
* Patients having vaginal delivery and LEA
* Singleton or Multiple pregnancy

Exclusion Criteria:

* under 18 years of age
* unwilling to provide written informed consent, or unable to follow the questions due to their mental state or language barriers.
* Patients who delivered via Cesarean section
* TOP/ IUFDs
* requiring instrumental deliveries- for example forceps or vacuum
* requiring to go to the OR postpartum for PPH or other reasons
* BMI at the time of delivery that falls in the super-morbidly obese category (BMI >55kg/m2)
* Preterm delivery (under 37 weeks of gestation)
* Patients who had inadvertent Dural Puncture during epidural placement
* Patients who had contraindicated or failed epidural anesthesia and required IV PCA for or during their delivery will also be excluded

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who deliver vaginally with neuraxial analgesia at Mount Sinai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Patient questionnaire | Following scheduled c-section delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be asked to rate their experience of having a vaginal delivery with neuraxial analgesia, in terms of satisfaction and their experience with any discomfort.
  Some questions are yes/no, some are on a scale from 1-10, where 1 = not at all and 10 = totally agree, and some are open-ended.
  The questionnaire will take approximately 10 minutes to complete.
Patient interview | Following scheduled c-section delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be interviewed in person by a member of the research team and asked open ended questions. Interviews will be recorded, transcribed and coded for themes.
  Responses are not reported on any scale. The interview will take approximately 30 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Nabecker, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No